CLINICAL TRIAL: NCT07275814
Title: A Multicenter, Randomized, Double-Blind, Positive-Controlled, Cross-Over Phase Ⅲ Clinical Trial Evaluating the Efficacy and Safety of HRS-9231 for Central Nervous System (CNS) Magnetic Resonance Imaging (MRI)
Brief Title: A Study of a Gadolinium-Based Contrast Agent (GBCA) for Adults Undergoing Magnetic Resonance Imaging (MRI) for Known or Highly Suspected Central Nervous System (CNS) Lesions
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Shengdi Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: HRS-9231-301
Record Dates: First submitted 2025-11-18; First posted 2025-12-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: For Contrast-enhanced Magnetic Resonance Imaging (MRI) of Central Nervous System (CNS) Lesions
MeSH Terms: interventions — gadobutrol; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gadobutrol + HRS-9231 Group (Experimental): HRS-9231 enhanced MRI then Gadobutrol enhanced MRI.
  Interventions: Drug: HRS-9231 Injection; Drug: Gadobutrol Injection; Device: Magnetic Resonance Imaging (MRI)
- HRS-9231 + Gadobutrol Group (Experimental): Gadobutrol enhanced MRI then HRS-9231 enhanced MRI.
  Interventions: Drug: HRS-9231 Injection; Drug: Gadobutrol Injection; Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: HRS-9231 Injection — HRS-9231 injection.
Drug: Gadobutrol Injection — Gadobutrol injection.
Device: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI).

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HRS-9231 for Central Nervous System (CNS) Magnetic Resonance Imaging (MRI); to demonstrate that, in patients requiring CNS MRI examinations, HRS-9231 is non-inferior to Gadobutrol in lesion visualization scores and show that, in patients requiring CNS MRI examinations, contrast-enhanced MRI with HRS-9231 is superior to unenhanced MRI in lesion visualization scores using the patients as their own controls; and to explore the population pharmacokinetic characteristics of HRS-9231 in CNS MRI subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form, willing to cooperate with the study, and comply with trial requirements.
2. Age ≥ 18 years, male or female.
3. Have at least one known or highly suspected CNS enhancement abnormality or lesion detected by imaging (e.g., CT and MRI) within 12 months prior to ICF signing.

Exclusion Criteria:

1. Clinically unstable condition or severe diseases that may affect trial results, such as inability to ensure imaging comparability or reliability of study parameters.
2. Severe renal impairment, defined as aGFR < 30 mL/min/1.73 m2.
3. Acute kidney injury, irrespective of eGFR levels.
4. Contraindications to MRI examinations or Gadobutrol, such as metallic implants ，pacemakers or claustrophobia.
5. History of severe allergies, including drugs, contrast agents, or other allergens.
6. Severe cardiovascular disease.
7. Female subjects who are pregnant or breastfeeding.
8. Other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
To compare the lesion visualization scores (border delineation) of HRS-9231-enhanced with gadobutrol-enhanced MRI. | Day 1 after procedure.
To compare the lesion visualization scores (internal morphology) of HRS-9231-enhanced with gadobutrol-enhanced MRI. | Day 1 after procedure.
To compare the lesion visualization scores (degree of contrast enhancement) of HRS-9231-enhanced with gadobutrol-enhanced MRI. | Day 1 after procedure.

SECONDARY OUTCOMES:
To compare the lesion visualization scores of HRS-9231-enhanced with unenhanced MRI. | Day 1 after procedure.
Number, size, and location of CNS lesions in MRI images after receiving HRS-9231. | Day 1 after procedure.
Number, size, and location of CNS lesions in MRI images after receiving gadobutrol. | Day 1 after procedure.
HRS-9231 plasma concentration. | Day 1 after procedure.
Population pharmacokinetic parameters - clearance. | Day 1 after procedure.
Population pharmacokinetic parameters - apparent volume of distribution. | Day 1 after procedure.
Overall diagnostic preference for CNS lesions on MRI images of HRS-9231 and gadobutrol. | Day 1 after procedure.
Diagnostic confidence of MRI images of HRS-9231 and gadobutrol. | Day 1 after procedure.
Technical adequacy of MRI images of HRS-9231 and gadobutrol. | Day 1 after procedure.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Henan Provincial People's Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: Undecided